CLINICAL TRIAL: NCT00424320
Title: Clinical Controlled Trial to Determinate the Role of Sodium Bicarbonate in the Prevention of Contrast-Induced Nephropathy in High-Risk Patients Undergoing to Diagnostic Coronariography and/or Percutaneous Coronary Intervention
Brief Title: Clinical Trial of Sodium Bicarbonate to Prevent Contrast-Induced Nephropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-001
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2007-01-19 (Estimated); Status verified 2007-01

CONDITIONS: Acute Kidney Failure
Keywords: Acute kidney failure; Contrast-induced nephropathy; Non-ionic contrast media; Ionic contrast media; Iopamidol; Percutaneous coronary intervention; Coronariography
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Bicarbonate

INTERVENTIONS:
Drug: Sodium bicarbonate

SUMMARY:
The purpose of this study is to determine whether sodium bicarbonate is effective in the prevention of sodium-induced nephropathy

DETAILED DESCRIPTION:
The use of contrast media is more frequent as new diagnostic and therapeutic procedures are developed. As a consequence, the occurrence of acute renal failure (ARF), also known as contrast-induced nephropathy, is more frequently seen after the realization of these procedures, representing about 10% of all in-hospital ARF. The importance of preventing this complication is related with its strong association with higher morbidity and mortality rates in patients who present it. A number of drugs and interventions have been studied for preventing contrast-induced nephropathy, including intravenous hydration with normal and hypotonic saline solutions, oral hydration, mannitol, diuretics, dopamine and its antagonists (fenoldopam), calcium antagonists, theophylline, N-acetylcysteine, natriuretic atrial peptide and hemodialysis after or during contrast media administration.

There is only one study in humans that demonstrates the utility of the sodium bicarbonate to prevent the contrast-induced nephropathy, showing a reduction in the incidence of this complication of about 13.6%. Although this result could seem convincing, its relevance has been questioned because the definition used by the authors as contrast-induced nephropathy was an increase of 25% from basal creatinine. Although when compared, the absolute differences between basal and after-procedure creatinines were not statistically significative, the sample size was small and the participants were low-risk patients to develop contrast-induced nephropathy. It is also important to note that the control group was hydrated with a dextrose 5% solution with 154 mEq of NaCl, although today's most accepted prevention therapy is intravenous hydration with normal saline solution.

Comparison: Hydration previously, during and afterwards contrast media administration with normal saline solution (0.9%), compared to hydration previous, during and afterwards contrast media administration with a solution made of normal saline and sodium bicarbonate.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Indication for coronariography and/or percutaneous coronary intervention
* Voluntary written consent for the realization of coronariography and/or percutaneous intervention and for the participation in this clinical trial
* A MEHRAN contrast-induced nephropathy score of six or more

Exclusion Criteria:

* Patients with chronic kidney failure requiring any kind of dialysis
* Patients unable to complete follow-up
* Multiple myeloma
* Exposure to contrast 48 hours prior to study
* Pregnancy
* Patients unable to give consent
* Already receiving sodium bicarbonate solutions
* Receiving contrast media other than non-ionic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-10; Study Completion 2007-01

PRIMARY OUTCOMES:
Contrast-induced nephropathy

SECONDARY OUTCOMES:
Hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Emma Miranda Malpica, PhD, Principal Investigator — Ignacio Chávez National Institute of Cardiology; Marco A Martínez Ríos, MD, FACC, Study Director — Ignacio Chávez National Institute of Cardiology; Jorge Gaspar Hernández, MD, Study Chair — Ignacio Chávez National Institute of Cardiology
Locations (2):
- Mexico (2):
  - ABC Medical Center, Mexico City, Mexico City (d.f.)
  - Ignacio Chávez National Institute of Cardiology, Mexico City, Mexico City (d.f:)

REFERENCES:
- [Background] Bagshaw SM, Ghali WA. Acetylcysteine for prevention of contrast-induced nephropathy after intravascular angiography: a systematic review and meta-analysis. BMC Med. 2004 Oct 22;2:38. doi: 10.1186/1741-7015-2-38. PMID 15500690
- [Background] Itoh Y, Yano T, Sendo T, Oishi R. Clinical and experimental evidence for prevention of acute renal failure induced by radiographic contrast media. J Pharmacol Sci. 2005 Apr;97(4):473-88. doi: 10.1254/jphs.crj05002x. Epub 2005 Apr 9. PMID 15821342
- [Background] Aspelin P. Nephrotoxicity and the role of contrast media. Radiat Med. 2004 Nov-Dec;22(6):377-8. No abstract available. PMID 15648451
- [Background] Mueller C, Seidensticker P, Buettner HJ, Perruchoud AP, Staub D, Christ A, Buerkle G. Incidence of contrast nephropathy in patients receiving comprehensive intravenous and oral hydration. Swiss Med Wkly. 2005 May 14;135(19-20):286-90. doi: 10.4414/smw.2005.10938. PMID 15986266
- [Background] Goldenberg I, Matetzky S. Nephropathy induced by contrast media: pathogenesis, risk factors and preventive strategies. CMAJ. 2005 May 24;172(11):1461-71. doi: 10.1503/cmaj.1040847. PMID 15911862
- [Background] Cavusoglu E, Chhabra S, Marmur JD, Kini A, Sharma SK. The prevention of contrast-induced nephropathy in patients undergoing percutaneous coronary intervention. Minerva Cardioangiol. 2004 Oct;52(5):419-32. PMID 15514576
- [Background] Rezkalla SH. Contrast nephropathy. Clin Med Res. 2003 Oct;1(4):301-4. doi: 10.3121/cmr.1.4.301. PMID 15931323
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Briguori C, Airoldi F, Morici N, Colombo A. New pharmacological protocols to prevent or reduce contrast media nephropathy. Minerva Cardioangiol. 2005 Feb;53(1):49-58. PMID 15788979
- See also: National Institute of Cardiology — http://www.cardiologia.org.mx